CLINICAL TRIAL: NCT04998630
Title: Comparison of Focused ESWT by Low and High Frequency for Patients With Myofascial Pain Syndrome: a Pilot Study
Brief Title: Comparison of Focused ESWT by Frequency for Patients With Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05-029
Record Dates: First submitted 2021-07-09; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Myofascial Pain Syndrome
Keywords: ESWT; myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (4Hz) (Experimental): ESWT frequency 4Hz washout period: 1 week
  Interventions: Device: Extracorporeal shockwave therapy
- B (8Hz) (Experimental): ESWT frequency 8Hz washout period: 1 week
  Interventions: Device: Extracorporeal shockwave therapy

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — Treatment Location: Painful Area Treatment intensity: 2000 pulses, low energy (0.08~0.28 mJ/m2) the degree to which the subject can tolerate

SUMMARY:
To investigate the efficacy and safety according to the frequency of focused ESWT in patients with myofascial pain syndrome.

DETAILED DESCRIPTION:
Myofascial pain syndrome is one of the common causes of musculoskeletal pain seen in clinical practice and is characterized by the presence of trigger points associated with sensitive areas such as taut bands of skeletal muscle. It may also be accompanied by referred pain, which is pain in other parts of the body. Although the pathophysiology and etiology of myofascial pain syndrome and trigger points are still unknown, there are reports that myofascial pain is a complex form of neuromuscular dysfunction caused by motor and sensory abnormalities involving both the peripheral nervous system and the central nervous system. Recently, it has been considered as a method of treatment for myofascial pain syndrome. In addition, although pain reduction and functional improvement of focused ESWT in patients with myofascial pain syndrome have been reported, related studies are lacking on the effect of focused ESWT according to the frequency difference. The purpose of the study is to examine the efficacy and safety of focused type ESWT frequency in patients with myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Those diagnosed with myofascial pain syndrome according to Simon's criteria
2. Pain is 4 points or more on the Numerical Rating Scale (NRS)

Exclusion Criteria:

1. Pain is due to trauma, fibromyalgia and neurological disorders including neuromyopathy, myelopathy, and stroke
2. If you have received injection treatment for trigger points within the last 2 months or have had surgery on the painful area within 1 year
3. If there is a high risk of bleeding due to severe coagulopathy, etc. or if you have recently had severe bleeding (except taking antiplatelet)
4. If you have a tumor, infection, kidney failure, severe liver disease, epilepsy, skin disease, or mental retardation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline NRS (numerical rating scale) at each time frame | baseline, immediately after primary treatment, 1 day after primary treatment, 3 day after primary treatment, immediately after secondary treatment, 1 day after secondary treatment, 3 day after secondary treatment
  Pain intensity (0-10, ordinal scale)

SECONDARY OUTCOMES:
Number of treatment-related adverse events as assessed by CTCAE v4.0 at each time frame | immediately after primary treatment, 1 day after primary treatment, 3 day after primary treatment, immediately after secondary treatment, 1 day after secondary treatment, 3 day after secondary treatment
  Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghoon Min, MD, PhD, Study Director — Department of Rehabilitation Medicine, CHA Bundang Medical Center, CHA University School of Medicine
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea